CLINICAL TRIAL: NCT02974309
Title: Extending Sleep to Improve Glycemic Control in Pediatric Type 1 Diabetes
Brief Title: Family Routines Enhancing Adolescent Diabetes by Optimizing Management
Acronym: FREADOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RDK110528A
Record Dates: First submitted 2016-04-27; First posted 2016-11-28 (Estimated); Last update posted 2024-11-27 (Actual); Status verified 2024-06

CONDITIONS: Type 1 Diabetes
Keywords: Youth; Diabetes Management; Sleep
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sleep Extension (Experimental): All youth in this condition are asked to extend their sleep to 10 hours or at least one hour, whichever is longer.
  Interventions: Behavioral: Sleep Extension
- Routine (Sham Comparator): All youth in this condition are asked to follow the routine that their clinical team has established.
  Interventions: Behavioral: Routine

INTERVENTIONS:
Behavioral: Sleep Extension — All youth in this condition are asked to extend their sleep to 10 hours or at least one hour, whichever is longer
  Arms: Sleep Extension
Behavioral: Routine — All youth in this condition are asked to follow the routines set by their clinical care team.
  Arms: Routine

SUMMARY:
A three month randomized study to examine the potential benefits of sleep extension in tandem with clinical trial on diabetes management in youth with type 1 diabetes.

DETAILED DESCRIPTION:
Type 1 Diabetes (T1DM) is one of the most common chronic medical conditions that occur in children. More than two-thirds of these young patients struggle to maintain optimal glycemic control. On a seemingly unrelated front, insufficient sleep has become a public health crisis as less than 30% of youth achieve the recommended number of hours on school nights. Prior research has supported that sleep disturbances contribute to elevated glucose levels and have a significant impact on memory, attention, and planning. These skills are essential to effective diabetes management. Despite the link between sleep and diabetes, no research has examined the benefits of an intervention to help these youth achieve a healthy sleep duration. To that end, our primary objective is to determine the effect of sleep extension on glycemic control and psychosocial functioning. Our secondary objective is to determine mediators and moderators of effect. The central hypothesis is that an increase in sleep duration will lower glucose levels and improve behavioral ratings (internalizing, externalizing, and classroom behaviors). Our primary study aims are to (1) Test if lengthening sleep improves glycemic control and psychosocial function in youth with T1DM; (2) Assess putative mechanisms for the effects of sleep extension on glucose and psychosocial function; and (3) Examine the possible moderating effect of pre-existing sleep parameters and sociodemographic variables that modify the impact of sleep extension. A secondary aim is exploratory to examine additional pre-selected mediators and moderators. In the proposed randomized study, up to 175 youth with T1DM will be assigned to a Sleep Extension or a supportive routines condition. The Sleep Extension lengthens youth's time in bed to allow for a healthy sleep duration on a consistent basis, whereas the supportive routines condition reinforces daytime and nighttime activities. We will test the impact of sleep extension on key indices of glycemic control (average glucose levels and % time hyperglycemia using continuous glucose monitors and HbA1C) as well as putative mechanisms of effect (e.g., heart rate variability and salivary cortisol levels) and participant characteristics that might mitigate the benefits of sleep extension (e.g., sleep-disordered breathing, adherence, and SES). Once our aims are achieved and a causal link is established, the proposed Sleep Extension intervention will advance knowledge about the role of sleep in diabetes management and provide a beneficial intervention to help youth with T1DM.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes

Exclusion Criteria:

* neurological, developmental, or psychiatric condition that in the opinion of the PI would significantly interfere with sleep or participation
* not hospitalized within the previous month prior to enrollment

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 115 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
HbA1c | 3 months
  A measure of glucose control

SECONDARY OUTCOMES:
Glucose Levels via continuous glucose monitor | 1 and 3 months
  Glucose levels will be measured at regular intervals using a subcutaneous continuous glucose monitor
Sleep Duration | 3 months
  Sleep duration will be measured using a combination of wrist actigraphy and polysomnography data.

OTHER OUTCOMES:
Diabetes Self-Management | 1 and 3 months
  Diabetes self-management and care activities will be assessed using the Diabetes Self-Management Profile for Flexible Regimes, Self- and Parent-proxy reports
Adherence to Diabetes Management | 1 and 3 months
  Adherence to diabetes management will be measured using the average daily manual glucose measurements from a personal glucometer (i.e. finger sticks)
Polysomnographic Sleep Architecture | 1 and 3 months
  Sleep architecture will be measured as percent time spent sleeping in the different stages of sleep (NREM 1, 2, 3, REM) using an in-home polysomnography system.
Quality of Life | 1 and 3 months
  Quality of Life will be measured using an aggregate of the Pediatric Quality of Life Inventory (PedsQL) Core 4.0 and Diabetes 3.2 modules.
Cortisol | 1 and 3 months
  Morning and evening Cortisol levels will be measured using a saliva collection device

CONTACTS AND LOCATIONS:
Overall Officials: Michelle M Perfect, PhD, Principal Investigator — UA College of Education
Locations (1):
- Pediatric Endocrinology Clinic, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon request.